CLINICAL TRIAL: NCT06019793
Title: Electrophysiological Recordings from Deep Brain Stimulation Electrodes for Pain
Acronym: EPR Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-500-326-30-06
Record Dates: First submitted 2023-08-22; First posted 2023-08-31 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- DBS for Chronic Pain (Experimental)
  Interventions: Device: DBS for Chronic Pain

INTERVENTIONS:
Device: DBS for Chronic Pain — Participants ill receive deep brain stimulation to relieve their chronic pain symptoms.

SUMMARY:
Over the last 30 years, deep brain stimulation (DBS) has allowed tens of thousands of patients to receive relief of neurological symptoms that were refractory to standard medical treatment. Furthermore, by providing a rare window into the electrophysiological activity of the awake, human brain, DBS has facilitated invaluable advances in scientific understanding. These advances have then, in turn, allowed for further therapies to be developed for an ever growing population of patients that benefit from DBS therapy. This study hopes to add to this growing body of knowledge by implanting leads within, and recording from, the sensory thalamus and periaqueductal gray (PAG) in patients with chronic pain. Specifically, we hope to establish the long-term safety of DBS leads within the periaqueductal gray and sensory thalamus for the treatment of chronic pain. Furthermore, by recording from the electrodes of DBS patients implanted for treatment of their chronic pain, we hope to understand how the pain network responds to sensory stimuli and how DBS changes this response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have intractable pain, as defined by: chronic (>1 year), severe (VAS score > 6/10), and persistent (not responsive to medication or relevant surgical options) without cognitive impairment or comorbidities affecting surgical risk.
2. Patients that have been medically cleared for DBS surgery by the consensus committee.
3. Not exhibiting significant distress, anxiety, or psychological disturbance that may be worsened due to externalized leads or potential complications or by study recording or tasks.
4. Motorically and cognitively capable of completing evaluations and consent.
5. Motorically and cognitively capable of participating in the study's computer-based tasks.
6. Informed consent signed by the subject.
7. Patient age between 22 to 75 years old.

Exclusion Criteria:

1. Patients that are not a candidate for DBS. This may occur for example, if they are unable to properly operate the neurostimulator. Also, several medical procedures and studies are not compatible with DBS. These include diathermy, transcranial magnetic stimulation, MRI procedures using radio-frequency coils, electroconvulsive therapy. Patients are receiving these treatments or plan to receive them in the future will not be eligible. Also, the safety of DBS has not been established for patients with a previous surgical ablation, dementia, coagulopathies, moderate to severe depression, or patients who are pregnant. Patients with these conditions will also not be eligible. Finally, DBS may be affected by or may affect other medical devices including cardiac pacemakers/defibrillator, ultrasonic equipment, radiation therapy, and incomplete (abandoned) prior DBS systems. Patients with these conditions/devices will not be eligible for the study.
2. Subjects who have pain that is not severe enough to be considered for DBS: shorter than 1 year duration, VAS score < 6/10), responsive to medication or relevant surgical options.
3. Subjects deemed to have a psychiatric illness that would potentially interfere or cause undue stress during the awake implantation surgery, the 1-3 week stimulation trial period, or the long term care of the DBS system are ineligible to undergo the DBS implantation procedure and thus would not be able to participate in this trial.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of DBS for Chronic Pain as Assessed by Incidence of Treatment-Related Adverse Events | 2 years

SECONDARY OUTCOMES:
Localized Brain Activity as Measured by Changes in LFP Activity in Relation to DBS | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No